CLINICAL TRIAL: NCT03444701
Title: A Phase 1 Study of E7130 in Subjects With Solid Tumor
Brief Title: A Study of E7130 in Participants With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: E7130-J081-101
Record Dates: First submitted 2018-02-04; First posted 2018-02-23 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumors
Keywords: Solid tumors; Squamous cell carcinoma of the head and neck; Urothelial carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Transitional Cell

STUDY DESIGN:
Intervention Model Description: This is a Phase 1 study of E7130 in participants with solid tumors. This study will be conducted in 2 parts (Part 1 and Part 2). Part 1 will be the dose escalation portion of this study, conducted to assess dose-limiting toxicity (DLT) and to determine the maximum tolerated dose (MTD) in participants with solid tumors. The dosage and the duration of the treatment cycle in Part 2 will be determined based on the data from Part 1. Part 2 will be comprised of cohort expansions to further characterize the safety and tolerability of E7130.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E7130 (2-Week Regimen) (Experimental): Part 1 (Cycle 1; 28 days): The first cohort of 3 participants will receive 25 micrograms per meters squared (μg/m^2) of E7130, on Day 1 and Day 15 as an intravenous infusion. If a drug-related Grade 2 or higher toxicity excluding clinically insignificant events is not observed in the initial cohort, dose-limiting toxicities (DLTs) will be evaluated in successive dose levels with single participants until such a toxicity is observed. Once the maximum tolerated dose (MTD) will be determined. Part 2: Participants with squamous cell carcinoma of the head and neck and urothelial carcinoma will be evaluated at the dose level determined in Part 1 in a 2-week or in a 3-week regimen based on the evaluations in Part 1.
  Interventions: Drug: E7130
- E7130 (3-Week Regimen) (Experimental): Part 1 (Cycle 1; 21 days): On Day 1, participants will receive E7130 at (-1) a lower dose than the dose at which the first DLT was observed in the 2-week regimen. Once the MTD will be determined. Part 2: Participants with squamous cell carcinoma of the head and neck and urothelial carcinoma will be evaluated at the dose level determined in Part 1 in a 3-week or in a 2-week regimen based on the evaluations in Part 1.
  Interventions: Drug: E7130

INTERVENTIONS:
Drug: E7130 — Starting dose of 25 μg/m^2 on Day 1 and Day 15 of Cycle 1.
  Arms: E7130 (2-Week Regimen)
Drug: E7130 — Starting dose is lower than one at which the first DLT was observed in the 2-week regimen administered on Day 1 of Cycle 1.
  Arms: E7130 (3-Week Regimen)

SUMMARY:
The primary objective of this study is to evaluate the tolerability and safety profile of E7130 in participants with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have provided voluntary written consent for participation in this clinical study
* Participants to whom the rules for complying with this clinical study have been adequately explained, and who intend to and can comply with these rules
* Participants aged greater than or equal to (>=) 20 years at the time of informed consent
* Participants with adequate function of major organs
* Participants with Performance Status score of 0 to 1 established by the Eastern Cooperative Oncology Group (ECOG)
* Participants who are expected to survive for 3 months or longer after starting administration of the investigational drug
* Washout period required from the end of prior treatment to the first administration of study drug
* Participants who agree to submit blood samples prior and during study treatment for progressive disease (PD) markers.

Inclusion Criteria (Part 2 only):

* Measurable disease meeting the following criteria:

  1. At least 1 lesion of >=1.0 centimeter (cm) in the longest diameter for a non-lymph node or >=1.5 cm in the short-axis diameter for a lymph node that is serially measurable according to response evaluation criteria in solid tumours (RECIST) 1.1 using computerized tomography/magnetic resonance imaging (CT/MRI).
  2. Lesions that have had external beam radiotherapy (EBRT) or locoregional therapies such as radiofrequency (RF) ablation must show evidence of progressive disease to be deemed a target lesion.

     Exclusion Criteria:
* Medical history of clinically significant cardiovascular impairment
* Serious concomitant systemic infection requiring medical treatment (including bacterial infection and fungal infection)
* Participants who test positive for human immunodeficiency virus (HIV antibody)
* Active viral hepatitis (B or C) as demonstrated by positive serology or requiring treatment hepatitis B surface antigen (HBsAg), anti-hepatitis B surface antibody (anti-HBs)/hepatitis B core antibody (HBcAb) and anti-hepatitis C virus (HCV) antibody test.
* Effusion requiring drainage
* Participants whose toxicity of previous treatment has not recovered to Grade 1 or lower (except for alopecia and hemoglobin)
* Other active malignancy
* Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin [ß-hCG] or human chorionic gonadotropin [hCG]).
* Women of childbearing potential or men of impregnate potential who don't agree that both the participant and his/her partner will use a medically effective method for contraception during the study and after study drug discontinuation (male; 90 days, female; 60 days)
* Known intolerance to the study drug or any of the excipients
* Any medical or other condition that in the opinion of the investigator(s) would preclude the participant's participation in the study
* Scheduled for surgery during the study
* Diagnosed with meningeal carcinomatosis
* Participants with brain or subdural metastases are not eligible.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of participants assigned to the every 2 weeks regimen with dose-limiting toxicities (DLTs) | Cycle 1 (28 days)
  DLTs are defined as study drug related adverse events (AEs). Toxicity will be evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03 (NCI CTCAE 4.03).
Part 1: Number of participants assigned to the every 3 weeks regimen with DLTs | Cycle 1 (21 days)
  DLTs are defined as study drug related AEs. Toxicity will be evaluated according to NCI CTCAE 4.03.
Part 1 and Part 2: Number of participants with adverse events (AEs) | Up to approximately 83 months
Part 1 and Part 2: Number of participants with any clinically significant clinical laboratory test value | Up to approximately 83 months
  Clinical significance will be determined by the Investigator.
Part 1 and Part 2: Number of participants with any clinically significant vital sign value | Up to approximately 83 months
  Clinical significance will be determined by the Investigator.
Part 1 and Part 2: Change from Baseline in arterial oxygen saturation | Baseline; Up to approximately 83 months
Part 1 and Part 2: Change from Baseline in body weight | Baseline; Up to approximately 83 months
Part 1 and Part 2: Number of participants with any clinically significant 12-lead electrocardiogram (ECG) value | Up to approximately 83 months
Part 1 and Part 2: Change from Baseline in the performance status (PS) score established by the Eastern Cooperative Oncology Group (ECOG) | Baseline; Up to approximately 83 months

SECONDARY OUTCOMES:
Part 1: Maximum Tolerated Dose (MTD) of E7130 | Cycle 1 and Cycle 2 (56 days [every 2 weeks regimen] [each Cycle length = 28 days], 42 days [every 3 weeks regimen] [each Cycle length = 21 days])
  The MTD will be selected as the dose with the smallest difference between the target DLT rate of 25% and an estimate of DLT rate based on the posterior distribution of DLT rate for each dose.
Part 1: Maximum observed plasma concentration (Cmax) of E7130 | Bi-weekly: Cycles 1-2 Days 1 and 15: 0-168 hours post-infusion (each Cycle length=28 days); Tri-weekly: Cycles 1-2 Day 1: 0-336 hours post-infusion (each Cycle length=21 days)
  Cmax is the maximum observed concentration of E7130 after administration of the drug.
Part 1: Time to reach maximum plasma concentration (Tmax) of E7130 | Bi-weekly: Cycles 1-2 Days 1 and 15: 0-168 hours post-infusion (each Cycle length=28 days); Tri-weekly: Cycles 1-2 Day 1: 0-336 hours post-infusion (each Cycle length=21 days)
  Tmax is the time at which the highest drug concentration occurs.
Part 1: Area under the plasma concentration time curve (AUC) from time 0 to infinity | Bi-weekly: Cycles 1-2 Days 1 and 15: 0-168 hours post-infusion (each Cycle length=28 days); Tri-weekly: Cycles 1-2 Day 1: 0-336 hours post-infusion (each Cycle length=21 days)
Part 1: Terminal elimination phase half-life (t1/2) of E7130 | Bi-weekly: Cycles 1-2 Days 1 and 15: 0-168 hours post-infusion (each Cycle length=28 days); Tri-weekly: Cycles 1-2 Day 1: 0-336 hours post-infusion (each Cycle length=21 days)
Part 1: Total clearance of E7130 | Bi-weekly: Cycles 1-2 Days 1 and 15: 0-168 hours post-infusion (each Cycle length=28 days); Tri-weekly: Cycles 1-2 Day 1: 0-336 hours post-infusion (each Cycle length=21 days)
Part 1: Volume of distribution (Vd) | Bi-weekly: Cycles 1-2 Days 1 and 15: 0-168 hours post-infusion (each Cycle length=28 days); Tri-weekly: Cycles 1-2 Day 1: 0-336 hours post-infusion (each Cycle length=21 days)
Part 1 and Part 2: Recommended dose for future studies | Up to approximately 83 months
  The recommended dose will be determined based on the on the MTD, the optimal biologic dose, and efficacy/safety/pharmacokinetic/pharmacodynamic data in Part 1 and Part 2.
Part 1 and Part 2: Number of participants with advanced solid tumors with anti-tumor activity | Up to approximately 83 months
Part 1 and Part 2: Best Overall Response (BOR) | Up to approximately 83 months
  The BOR will be based on Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. BOR is defined as complete response (CR), partial response (PR), stable disease (SD), progression of disease (PD), and not evaluable (NE), where SD has to be achieved at ≥5 weeks after the first dose.
Part 1 and Part 2: Objective Response Rate (ORR) | Up to approximately 83 months
  The ORR is defined as the percentage of participants with a BOR of CR or PR.
Part 1 and Part 2: Disease Control Rate (DCR) | Up to approximately 83 months
  DCR is defined as the percentage of participants with a BOR of CR, PR, or SD.
Part 1 and Part 2: Clinical Benefit Rate (CBR) | Up to approximately 83 months
  The CBR is defined as the percentage of participants with a BOR of CR, PR, or durable SD (duration of SD ≥23 weeks).
Part 2: Progression-free survival (PFS) | Up to approximately 83 months
  PFS is defined as the time from the date of the first dose to the first documented date of the event (disease progression or death from any cause, whichever occurs first).
Part 2: Overall Survival (OS) | Up to approximately 83 months
  OS is defined as the time from the date of the first dose to the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (9):
- Japan (9):
  - Eisai Trial Site 9, Nagoya, Aichi-ken
  - Eisai Trial Site 1, Kashiwa, Chiba
  - Eisai Trial Site 6, Kashiwa, Chiba
  - Eisai Trial Site 8, Sapporo, Hokkaido
  - Eisai Trial Site 4, Sendai, Miyagi
  - Eisai Trial Site 5, Chuo-ku, Osaka
  - Eisai Trial Site 7, Bunkyo-ku, Tokyo
  - Eisai Trial Site 3, Chuo-ku, Tokyo
  - Eisai Trial Site 2, Koto-ku, Tokyo

REFERENCES:
- [Derived] Doi T, Matsubara N, Naito Y, Kuboki Y, Harano K, Ono M, Urasaki T, Ohmoto A, Kawanai T, Hisai T, Ikezawa H, Shiba S, Ito K, Semba T, Asano O, Takahashi S. First-in-human study of E7130 (a tumor microenvironment-ameliorating microtubule inhibitor) in patients with advanced solid tumors: Primary results of the dose-escalation part. Cancer. 2023 Aug 1;129(15):2348-2359. doi: 10.1002/cncr.34788. Epub 2023 Apr 20. PMID 37080942